CLINICAL TRIAL: NCT06871033
Title: Comparison Between Ketamine and Neostigmine As Adjuvants to Bupivacaine in Ultrasound-Guided Transversus Abdominis Plane Block in Caesarean Section
Brief Title: Ketamine Versus Neostigmine in Ultrasound-Guided Transversus Abdominis Plane Block in Caesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0201931
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-12

CONDITIONS: Caesarian Section; Postoperative Pain
Keywords: Ketamine; Neostigmine; TAP block; Caesarian section; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Neostigmine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP block with Ketamine (Active Comparator): 40 patients will receive postoperative TAP block with 20 ml 0.25% plain bupivacaine (10ml 0.5% bupivacaine added to 10ml normal saline) and 0.5 mg/kg ketamine for each side
  Interventions: Drug: TAP block with Ketamine
- TAP block with Neostigmine (Experimental): 40 patients will receive postoperative TAP block with 20ml 0.25% plain bupivacaine (10ml 0.5% bupivacaine added to 10ml normal saline) and 500 microgram neostigmine for each side.
  Interventions: Drug: TAP block with neostigmine

INTERVENTIONS:
Drug: TAP block with neostigmine — 40 patients will receive postoperative TAP block with 20ml 0.25% plain bupivacaine (10ml 0.5% bupivacaine added to 10ml normal saline) and 500 microgram neostigmine for each side.
  Arms: TAP block with Neostigmine
Drug: TAP block with Ketamine — 40 patients will receive postoperative TAP block with 20 ml 0.25% plain bupivacaine (10ml 0.5% bupivacaine added to 10ml normal saline) and 0.5 mg/kg ketamine for each side.
  Arms: TAP block with Ketamine

SUMMARY:
The current study investigates the efficacy and safety of ketamine and neostigmine as adjuvants in transversus abdominis plane blocks for Cesarean sections. The study participants arerandomized into two groups, each receiving either ketamine or neostigmine alongside plain bupivacaine. Various parameters, including pain intensity, intraoperative and postoperative hemodynamics, rescue analgesia requirements, patient satisfaction, and postoperative complications, are evaluated and compared between the two groups.

DETAILED DESCRIPTION:
A prospective, experimental double-blind control study will be conducted in Alexandria Main University Hospital after approval of the medical ethics committee of the Alexandria Faculty of Medicine and a written formal consent will be signed out from patients or their relatives. Patients will be double-blinded randomized into two equal groups (40 patients each) after receiving spinal anesthesia with 12.5 mg of 0.5% hyperbaric bupivacaine:

* Group 1: 40 patients received postoperative TAP block with 20 ml 0.25% plain bupivacaine (10ml 0.5% bupivacaine added to 10ml normal saline) and 0.5 mg/kg ketamine for each side.
* Group 2: 40 patients received postoperative TAP block with 20ml 0.25% plain bupivacaine (10ml 0.5% bupivacaine added to 10ml normal saline) and 500 microgram neostigmine for each side.

Preoperative assessment and preparation:

* Proper history taking.
* Complete clinical examination.
* Routine laboratory investigations.
* The technique of anaesthesia and visual analog score (VAS) will be explained to patients. The VAS score is a simple and commonly used method to measure pain intensity. It involves a horizontal line, usually 10 centimeters long, with one end representing "no pain" and the other end representing "worst pain imaginable." Patients will be asked to mark a point on the line that corresponds to their current pain level. This will help to understand the severity of pain and to determine the appropriate pain management strategies.
* Additionally, the difference between somatic or parietal pain and visceral pain will be explained to patients. Somatic or parietal pain arises from the outer layers of the body, such as the skin, muscles, and tissues. It is typically well-localized and sharp in nature, and increased with movement. In contrast, visceral pain originates from internal organs and is often described as dull, aching, or cramp-like that does not increase with movement. By understanding these distinctions, patients can better communicate their pain experiences.

Patient preparation:

The patients receive:

* Oral Famotidine 40 mg at night before the day of surgery.
* Ondansetron 4 mg IV immediately before surgery. Monitoring A multichannel monitor (Dräger, Vista 120) will be connected to the patient to display continuous electrocardiography monitoring for heart rate (beat/min) and detection of dysrhythmias, non-invasive arterial blood pressure (NIBP), pulse oxygen saturation (SpO2). Anaesthetic technique All patients undergoing elective CS surgery will receive spinal anaesthesia as the primary anaesthetic technique. Following the completion of the CS surgery, a Transversus Abdominis Plane (TAP) block will be performed to enhance postoperative pain management. Patient will be positioned supine on the operating table and the abdomen will be prepared and draped in a sterile manner to maintain aseptic conditions. Strict sterile techniques will be followed, including the use of sterile gloves, drapes, and local antiseptic solution for skin preparation. The ultrasound probe will be covered with a sterile sheath or barrier to ensure asepsis.

The TAP block will be performed using Sonosite M-turbo ultrasound with high-frequency (10-15 MHz) linear transducer. The skin will be disinfected with antiseptic solution. A linear transducer will be placed in the axial plane on the midaxillary line between the subcostal margin and the iliac crest. The three layers of abdominal wall muscles will be visualized: external and internal oblique as well as the transversus abdominis muscles. The target is the fascial plane between the internal oblique and the transversus abdominis muscles. The needle will be inserted in the anterior axillary line, and the needle tip will be advanced until it reaches the fascial plane then 20 ml of 0.25% plain bupivacaine and 0.5 mg/kg ketamine will be injected in the first group and 50 microgram neostigmine in the second group under repeated aspiration for every 5 milliliters separating the plane between the internal oblique and transversus abdominis muscles with increased radiotranslucency approximately in the midaxillary line. The identical technique will be repeated on the opposite side.

Over the next 24 hours, all patients received 1 g of paracetamol IV every 8 hour as a part of multimodal analgesia. Measurements

The following parameters will be measured in every patient in the study:

1. Vital signs Including heart rate (bpm), and mean arterial blood pressure (mmHg). All previous parameters will be continuously monitored and recorded before starting the surgery, intraoperatively and postoperatively after giving TAP block with adjuvants, at 2, 4, 6, 12, 18, and 24 hours postoperative.
2. Pain scoring The visual analog scale (VAS) will be recorded intraoperatively and at 2 hr., 4 hr., 6 hr., 12 hr., 18hr., and 24 hr. postoperatively. The rescue analgesia (nalbuphine 6 mg IV) will be used when VAS score ≥ 4.
3. Duration of analgesia (hours) Duration of analgesia defined as the time interval after start of the technique till the first need of rescue analgesic (nalbuphine 6 mg IV).
4. Total dose of rescue analgesia (mg) Cumulative use of opioid (nalbuphine) in 24 hours.
5. Patient satisfaction Patient satisfaction with the pain control will be assessed on a four-point scale as: Excellent, Good, Fair and Poor.
6. Complications Any post-operative complication occurred at any time in the 24 hours of the study will be recorded and analyzed accordingly:

   * Haemodynamic instability.
   * Haematoma at the site of injection.

ELIGIBILITY:
Inclusion criteria

* ASA physical status I or II patients.
* Patients undergoing elective CS. Exclusion criteria
* Patients undergoing emergent CS.
* Patient refusal.
* Allergy to local anaesthesia or any additive drug.
* Coagulopathy.
* Body mass index > 35.
* Peripheral neuropathy or chronic pain syndrome.
* Localized infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain score | Intraoperatively and at 2 hr., 4 hr., 6 hr., 12 hr., 18hr., and 24 hr. postoperatively
  Change From Baseline in Pain Scores on the Visual Analog Scale

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours postoperative
  Patient satisfaction with the pain control will be assessed on a four-point scale as: Excellent, Good, Fair and Poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Alexandria Governorate, Egypt